CLINICAL TRIAL: NCT06682169
Title: A Randomized, Open Label, Positive Controlled, Multicenter Phase III Clinical Trial Evaluating the Efficacy and Safety of the Selected Regimen of Rovadicitinib in Moderate to Severe Chronic Graft-versus-host Disease in Third Line and Beyond
Brief Title: Evaluation of Rovadicitinib Compared to the Protocol Selected by Researchers in Third Line and Subsequent Studies of Moderate to Severe Chronic Graft-versus-host Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-III-01
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Graft-versus-host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Imatinib Mesylate; Methotrexate; Mycophenolic Acid; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rovadicitinib (Experimental): Rovadicitinib: 10mg, taken orally on an empty stomach twice a day, with a minimum interval of 8 hours between each dose, and an optimal interval of 12 hours. Every 28 days is a treatment cycle.
  Interventions: Drug: Rovadicitinib
- Imatinib or Methotrexate or Mycophenolate or Rituximab (Active Comparator): Methotrexate tablets: 10mg, orally, once a week or 5mg, orally, twice a week.
  Metoprolol ester: 250mg-500mg, bid, orally.
  Imatinib: 100-400mg, qd, oral.
  Rituximab: 375mg/m2, administered intravenously once a week for 4 consecutive weeks.
  Interventions: Drug: Imatinib; Drug: Methotrexate; Drug: Mycophenolate mofetil; Drug: Rituximab

INTERVENTIONS:
Drug: Rovadicitinib — Rovadicitinib is an inhibitor of Janus associated kinases (JAK) family and Rho associated kinases (ROCK). It can inhibit the sustained abnormal activation of the Janus kinase (JAK) signal transducer and activator of transcription (JAK-STAT) pathway and also inhibit Rho associated kinase 2 (ROCK2). The JAK 1-JAK 2 signaling pathway is a key step in causing inflammation and tissue damage in acute and chronic graft-versus-host disease.
  Arms: Rovadicitinib
Drug: Imatinib — Imatinib tyrosine kinase inhibitor is a small molecule protein kinase inhibitor that has the ability to block one or more protein kinases. Clinically used for the treatment of chronic myeloid leukemia and malignant gastrointestinal stromal tumors.
  Arms: Imatinib or Methotrexate or Mycophenolate or Rituximab
Drug: Methotrexate — Methotrexate is an organic compound, mainly used as an anti folate anti-tumor drug. It inhibits the synthesis of tumor cells by inhibiting dihydrofolate reductase, thereby inhibiting the growth and reproduction of tumor cells.
  Arms: Imatinib or Methotrexate or Mycophenolate or Rituximab
Drug: Mycophenolate mofetil — Metoprolol ester is an organic compound mainly used as an immunosuppressant
  Arms: Imatinib or Methotrexate or Mycophenolate or Rituximab
Drug: Rituximab — Rituximab activates antibody dependent cell-mediated phagocytosis and complement dependent cytotoxicity by binding to cluster of differentiation 20 (CD20) antigen, clearing malignant B cells expressing CD20 and achieving therapeutic goals.
  Arms: Imatinib or Methotrexate or Mycophenolate or Rituximab

SUMMARY:
The aim of this study is to demonstrate that in subjects with moderate to severe chronic graft-versus-host disease in the third line and beyond, the use of rosuvastatin compared to the protocol chosen by the researchers can significantly improve the objective response rate of subjects at week 24.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years old; Karnofsky (KPS) ≥ 60 points; Expected survival period exceeding 6 months;
* Previously received allogeneic hematopoietic stem cell transplantation;
* According to NIH standards, the clinical diagnosis is moderate to severe cGVHD；
* Previously received systematic treatment for cGVHD with 2-5 lines;
* Stable dosage of corticosteroids and other immunosuppressants received within 2 weeks prior to screening;
* The main organ functions well;
* Starting from Day 1 after enrollment in the control group of this study, participants must receive one of the drugs specified in the study protocol;
* Female participants of childbearing age should agree to use contraceptive measures (such as intrauterine devices, birth control pills, or condoms) during the study period and for 6 months after the end of the study; Serum pregnancy test negative within 7 days prior to enrollment in the study, and must be a non lactating subject; Male participants should agree to use contraceptive measures during the study period and within 6 months after the end of the study period;
* Subjects voluntarily joined this study, signed informed consent, and had good compliance.

Exclusion Criteria:

* Has experienced or currently suffers from other malignant tumors within the past 3 years;
* Known or suspected active aGVHD；
* Individuals with interstitial pneumonia, non infectious pneumonia, uncontrolled active infections, or infections requiring systematic treatment within the first 7 days of randomization, except for those deemed suitable for inclusion by the researchers;
* The occurrence and progression of other underlying diseases include post transplant lymphoid tissue proliferative diseases and recurrence of primary malignant hematological diseases;
* Random failure of allogeneic hematopoietic stem cell transplantation within the first 6 months or having received 2 allogeneic hematopoietic stem cell transplants in the past;
* Used JAK inhibitors, Bruton's tyrosine kinase (BTK) inhibitors, etc. within the first 2 weeks of randomization;
* There are multiple factors that can affect oral medication, such as inability to swallow, intestinal obstruction, etc;
* Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
* Subjects with any severe and/or uncontrolled illnesses;
* Individuals who are allergic to research drugs or their components;
* Participated in other clinical trials within the first 4 weeks of randomization;
* According to the researcher's judgment, there are accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are deemed unsuitable for inclusion due to other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate in the 24th week (ORR) | Week 24
  Researchers evaluated each organ according to the consensus criteria of the NIH 2014 conference, and at week 24, the percentage of subjects with complete response (CR) or partial response (PR) in all assessable organs was determined.

SECONDARY OUTCOMES:
Best Objective Response Rate (BOR) | Week 24
  The best therapeutic effect among all therapeutic outcomes
Duration of Relief (DOR) | Through study completion, an average of 2 year
  The duration of symptom relief for patients after receiving treatment
Improvement in Lee cGVHD symptom score of subjects in week 24 | Week 24
  The Lee cGVHD Symptom Score is a tool used to assess the severity of symptoms in chronic graft-versus-host disease (cGVHD), ranging from 0 to 4 points, with a maximum total score of 16 points. The higher the score, the more severe the cGVHD symptoms.
Failure free survival (FFS) | Weeks 2, 4, 8, 16, 36, 48, 60, 72, 84, 96
  The time from the start of treatment to the occurrence of disease progression or death for any reason in the patient
Primary disease recurrence rate (MR) | Weeks 8, 16,24， 36, 48
  The probability of recurrence of the patient's disease within a certain period of time.
Non-Relapse Mortality (NRM) | Weeks 8, 16,24， 36, 48
  NRM was defined as death without recurrent or progressive disease
Overall survival (OS) | Through study completion, an average of 2 year
  From randomization to the time of death caused by any reason
Percentage of subjects whose daily glucocorticoid dose decreased | Week 24
  Percentage of subjects whose daily glucocorticoid dose decreased by ≥ 50% in week 24, and percentage of subjects who discontinued all glucocorticoids
Changes in the Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT) | Through study completion, an average of 2 year
  The FACT-BMT scale is a tool used to evaluate the quality of life (QOL) of patients after hematopoietic stem cell transplantation, the scale is filled out by the person closest to the patient, and each question has five possible answers on a scale of 0-4. Answer each question item based on the patient's actual situation in the past week, and mark the corresponding number with a "√"
Changes in 5-level EQ-5D (EQ-5D-5L) | Through study completion, an average of 2 year
  The scoring criteria of EQ-5D-5L scale include five dimensions: action ability, self-care ability, daily activity ability, pain or discomfort, anxiety or depression. After selecting a level for each dimension, a specific rating can be obtained. For example, if an individual chooses "slightly difficult" in terms of action ability, they will score 2 points on that dimension (from 0 to 5, where 0 indicates no difficulty and 5 indicates inability/very serious difficulty)
Adverse events (AE) | Through study completion, an average of 2 year
  The incidence and severity of adverse events (AE) and serious adverse events (SAE), as well as abnormal laboratory test indicators.
Cmax | Day 1, day 8 on cycle 1: 0.5 hour pre-dose, 0.5 hour after dose, day 1 cycle 2: 0.5 hour pre-dose, 2 hours after dose, day 1 cycle 4: 0.5 hour pre-dose, 3 hours after dose, day 1 cycle 6: 0.5 hour pre-dose, 4 hours after dose (28 days as a cycle)
  The maximum concentration of medication that enters the bloodstream after administration
Ctrough | Day 1, day 8 on cycle 1: 0.5 hour pre-dose, 0.5 hour after dose, day 1 cycle 2: 0.5 hour pre-dose, 2 hours after dose, day 1 cycle 4: 0.5 hour pre-dose, 3 hours after dose, day 1 cycle 6: 0.5 hour pre-dose, 4 hours after dose (28 days as a cycle)
  After multiple administrations, the blood drug concentration reaches a relatively stable state, which is called the steady-state concentration

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The 904 Hospital of the Joint Service Support Force of the People's Liberation Army of China, Lanzhou, Gansu
  - Guangzhou First People's Hospital The First People's Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical Hospital, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhenzhou, Henan
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tai'an City Central Hospital, Tai’an, Shandong
  - Shanghai Jiao Tong University School of Medicine，Renji Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Chinese Academy of Medical Sciences Hematology Hospital, Tianjin, Tianjin Municipality
  - The First Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang